CLINICAL TRIAL: NCT01365767
Title: Kontrast UltraLydsskanning af Tyndtarmen Hos Patienter Med Crohns Sygdom - et Pilotstudie. (Danish) Contrast Ultrasound of the Small Intestine in Patients With Crohns Disease - a Pilot Study (English)
Brief Title: Contrast Ultrasound of the Small Intestine in Patients With Crohns Disease
Acronym: KULT
Status: Completed | Type: Observational
Sponsor: Rune Wilkens (Other)
Responsible Party: Sponsor-Investigator, Rune Wilkens, MD, Regionshospitalet Silkeborg
Organization: Regionshospitalet Silkeborg (Other)
Other Study IDs: HGRWLBKULT1; 2010-024528-12 (EudraCT Number)
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Crohn Disease
Keywords: Crohn disease; Ultrasonography, contrast enhanced; Elasticity Imaging Techniques; Small intestine; Magnetic Resonance Imaging; CDAI; Calprotectin; IBD; Sonography
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Crohn Disease: Patients with Crohns Disease referred to referred to a Magnetic Resonance Imaging Scan.

SUMMARY:
The purpose of this study is to determine how relevant dynamic ultrasound scans using contrast agents (SonoVue) is in the diagnosis of Crohns disease in the small bowel, compared to dynamic Magnetic Resonance Imaging (MRI) of the small bowel.

DETAILED DESCRIPTION:
Crohns disease (CD) is a lifelong chronic Inflammatory Bowel Disease (IBD) normally with an early debut. It requires continuous evaluation with either endoscopy, Magnetic Resonance Imaging (MRI), Computed Tomography (CT) or Wireless Capsule Endoscopy (WCE). These methods are either expensive, invasive or with uses radiation. Therefore UltraSound (US), as a cheap, fast and well tolerated examination of the small bowel are tested against the the validated MRI examination of the small bowel. Both examinations are using intra venous (i.v.) contrast agents. Obtained results are compared to disease activity.

Hypothesis is, that dynamic US is comparable to dynamic MRI and therefore should be the first examination of choice in evaluating patients with CD.

This study is a pilot study only.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Crohns Disease
* 18 years old or older.
* Referred to a Magnetic Resonance Imaging scan of the small bowel

Exclusion Criteria:

* Contraindications to or not suitable of a Magnetic Resonance Imaging
* Liver transplant
* nursing og pregnancy
* Known Allergy of SonoVue
* Acute Myocardial infarction < 4 weeks
* Coronary angiography < 4 weeks
* Electrocardiogram changes < 4 weeks
* frequent and repetitive angina pectoris symptoms within the last week.
* Heartfailure
* serious arrhythmia
* right to left heart shunt
* Very high pulmonary artery pressure
* uncontrolled hypertension
* Adult respiratory distress syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated on Regional Hospital of Silkeborg.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Correlation between time-intensity curves of dynamic ultrasound and dynamic Magnetic Resonance Imaging | up to 1 week
  Time intesity curves are obtained using intra venous contrast agents during Magnetic Resonance Imaging scans and Ultrasound examination of the small bowel

SECONDARY OUTCOMES:
Correlation between elastography scans of Magnetic Resonance Imaging and Ultrasound of the small bowel | up to 1 week
Correlation between Doppler Score and Contrast Enhanced Ultrasound Score | up to 1 week
  Doppler score (Limberg score) and Contrast Enhanced Ultrasound score are obtained during the same scanning procedure
Correlation between greatest bowel wall thickness and disease activity measured in Ultrasound and Magnetic Resonance Imaging | up to 1 week
Correlation between Ultrasound score and Faeces Calprotectin | up to 2 months
Correlation between Crohns disease activity index and Ultrasound score | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Glerup, Study Chair — Region Hospital of Silkeborg; Rune Wilkens, Principal Investigator — Region Hospital of Silkeborg; Lars B. Hansen, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Medical department, Regional Hospital of Silkeborg, Silkeborg